CLINICAL TRIAL: NCT03272880
Title: Utilizing the Arts to Improve Health, Resilience, and Well-Being in Individuals With Cancer and Their Caregivers: A Feasibility Study
Brief Title: Utilizing the Arts to Improve Health, Resilience, and Well-Being Among Cancer Patients and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE14Z17
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Cancer
Keywords: Art Therapy; Music Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be a pre-post intervention observational study utilizing a mixed methods approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arts-based programming for cancer survivors and caregivers (Experimental): This is a 8-week, arts-based, health, resilience, and well-being program.
  Interventions: Behavioral: Arts-Based Programming

INTERVENTIONS:
Behavioral: Arts-Based Programming — This feasibility study includes educational components and an experiential components which are assessed with pre- and post-tests. The topics of these components include: Introduction to the Arts and Health; Music, Well-Being, and Resilience; Movement and Physical Activity; Art and Well-Being; Theater and Socialization; Art Appreciation and a Healthy Brain; and Summary/Integration of the Arts into Daily Lives. The impact of this program will be assessed with qualitative follow-up interviews.

SUMMARY:
The purpose of this study is to evaluate the impact of arts-based programming on health, well-being, and resilience. Patients who have cancer or are the caregivers of someone with cancer are being asked to take part in this study.

DETAILED DESCRIPTION:
Objective:

Primary:

To assess the feasibility and acceptability of arts-based programming for community-dwelling cancer survivors and caregivers. Feasibility and acceptability will be assessed based on:

1. Recruitment
2. Participation
3. Retention (drop-outs)
4. Satisfaction

Secondary:

To assess the participants' ability to:

1. Define goals and strategies using the contents of the program.
2. Implement the strategies in their daily activities in the short-term.
3. Continue to use these strategies after the program ends.

Exploratory:

To perform exploratory analyses on the impact of arts-based programming on health, resilience, and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in all program sessions
* Cognitively able to consent to participate
* Speaks, reads, and writes English
* Diagnosis of cancer or caregiver of someone with cancer

Exclusion Criteria:

* Severe visual or auditory impairment
* Severe and/or uncontrolled comorbidity precluding safe participation in a physical activity program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Feasibility: Number of participants recruited in the study | Up to 8 weeks after beginning of study
  Study will be feasible if recruitment goal is met with 10-20 participants enrolled
Feasibility: Average number of session attended by participants | Up to 8 weeks after beginning of study
  Study will be feasible if average number of session attended will be greater than or equal to 4
Percent of patients who drop out of study | Up to 8 weeks after beginning of study
  Study will be feasible if no more than 25% of patients drop out of study
Satisfaction Score | Up to 8 weeks after beginning of study
  Satisfaction will be high in post-test surveys

SECONDARY OUTCOMES:
Qualitative Impact of arts-based programming on health | Up to 3 weeks after final session (11 weeks from beginning of study)
  Impact of program on health described in phenomenological interviews
Qualitative Impact of arts based programming on resilience | Up to 3 weeks after final session (11 weeks from beginning of study)
  Impact of program on resilience described in phenomenological interviews
Qualitative Impact of arts based programming on well-being | Up to 3 weeks after final session (11 weeks from beginning of study)
  Impact of program on well-being described in phenomenological interviews

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Gallagher, MA, MT-BC, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States